CLINICAL TRIAL: NCT02445209
Title: Comparison of Efficacy and Frequency of Adverse Events of 1st Line Palliative Chemotherapy EOX and mDCF Regimens in Advanced HER2-negative Gastric Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Sebastian Ochenduszko, Sebastian Ochenduszko, MD PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JagiellonianU-01
Record Dates: First submitted 2015-04-30; First posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: HER2 Negative Gastric Cancer
Keywords: HER2-negative gastric and GEJ adenocarcinoma; first-line palliative chemotherapy; EOX; mDCF; efficacy; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EOX (Active Comparator): Epirubicin 50mg/m2 IV on day 1; Oxaliplatin 130mg/m2 IV on day 1; Capecitabine 625mg/m2/day PO BID days 1-21; Cycled every 21 days. Cycled every 3 weeks for a maximum of 8 cycles initially (24 weeks of treatment).
  Patients who experienced a long term response to the initial 8 cycles of EOX chemotherapy, could be rechallenged with the same regimen.
  Interventions: Other: EOX
- mDCF (Active Comparator): Docetaxel 40 mg/m2 IV od day 1; Leucovorin 400 mg/m2 IV on day 1; 5fluorouracyl 400 mg/m2 IV on day 1; 5fluorouracil 1000 mg/m2/d IV continuous infusion days 1-2; Cisplatin 40 mg/m2 IV on day 3; Cycled every 2 weeks for a maximum of 12 cycles initially (24 weeks of treatment).
  Patients who experienced a long term response to the initial 12 cycles of mDCF chemotherapy, could be rechallenged with the same regimen
  Interventions: Other: mDCF

INTERVENTIONS:
Other: EOX — combined chemotherapy regimen: epirubicin + oxaliplatin + capecitabine
  Arms: EOX
Other: mDCF — combined chemotherapy regimen: docetaxel + leucovorin + 5fluorouracil + cisplatin
  Arms: mDCF

SUMMARY:
The purpose of the study is to compare efficacy and safety of palliative chemotherapy EOX and mDCF regimens in the first-line treatment of patients with advanced HER2-negative gastric and gastroesophageal junction (GEJ) adenocarcinoma

DETAILED DESCRIPTION:
The main purposes: to determine the overall survival (OS) of patients who have locally advanced inoperable or metastatic HER2-negative gastric and gastroesophageal adenocarcinoma treated with first-line EOX (epirubicin + oxaliplatin + capecitabine) or mDCF (docetaxel + cisplatin + leucovorin + 5fluorouracil) palliative chemotherapy regimens

The secondary purposes: to determine safety (as assessed by adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.0) and the progression-free survival (PFS)

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* histologically confirmed inoperable locally advanced, recurrent, or metastatic adenocarcinoma of the stomach or gastro-oesophageal junction;
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2;
* adequate renal, hepatic, and hematologic function;
* measurable or nonmeasurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST). Patients with intraoperatively confirmed intraperitoneal metastases but without detectable disease in radiological studies were also eligible

Exclusion Criteria:

* HER2- positive tumors defined as either IHC 3+ or IHC 2+, the latter in combination with FISH+
* previous chemotherapy for metastatic or locally advanced disease
* surgery <3 weeks before the onset of the study treatment
* congestive heart failure
* significant dysphagia that would preclude oral administration of capecitabine
* concurrent malignant disease, except for adequately treated tumors with high likelihood of being cured (e.g. basal cell carcinoma of the skin, cervical cancer)
* clinical evidence of brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 years
  time from randomization until death from any cause

SECONDARY OUTCOMES:
Progression-free Survival | 3 years
  time from randomization to disease progression or death from any cause
Safety as assessed by adverse events according to CTCAE v4.0 | 3 years
  occurrence of adverse events according to CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Ochenduszko, M.D., PhD, Principal Investigator — Jagiellonian University

REFERENCES:
- [Background] Cunningham D, Starling N, Rao S, Iveson T, Nicolson M, Coxon F, Middleton G, Daniel F, Oates J, Norman AR; Upper Gastrointestinal Clinical Studies Group of the National Cancer Research Institute of the United Kingdom. Capecitabine and oxaliplatin for advanced esophagogastric cancer. N Engl J Med. 2008 Jan 3;358(1):36-46. doi: 10.1056/NEJMoa073149. PMID 18172173
- [Background] Shah MA, Stoller R, Shibata S, et al. Random assignment multicenter phase II study of modified docetaxel, cisplatin, fluorouracil (mDCF) versus DCF with growth factor support (GCSF) in metastatic gastroesophageal adenocarcinoma (GE). 2010 Gastrointestinal Cancers Symposium.
- [Derived] Ochenduszko S, Puskulluoglu M, Konopka K, Fijorek K, Urbanczyk K, Budzynski A, Matlok M, Lazar A, Sinczak-Kuta A, Pedziwiatr M, Krzemieniecki K. Comparison of efficacy and safety of first-line palliative chemotherapy with EOX and mDCF regimens in patients with locally advanced inoperable or metastatic HER2-negative gastric or gastroesophageal junction adenocarcinoma: a randomized phase 3 trial. Med Oncol. 2015 Oct;32(10):242. doi: 10.1007/s12032-015-0687-7. Epub 2015 Sep 9. PMID 26354521